CLINICAL TRIAL: NCT02893345
Title: Safe@Home: A Self-Management Program for Individuals With Traumatic Brain Injury and Their Families
Brief Title: Safe@Home: A Self-Management Program for Individuals With TBI and Their Families
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shepherd Center, Atlanta GA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 627-605210-2
Record Dates: First submitted 2016-08-25; First posted 2016-09-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Brain Injuries, Traumatic
Keywords: Self Care (Rehabilitation); Community Participation; Patient-Centered Outcomes Research; Informatics, Clinical
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safe@Home Intervention Group (Experimental): Participants receive: (1) computer-generated, personalized assessment of abilities, risk, and recommended next steps; (2) 2 person-family education visits to develop a shared understanding of client strengths and risks, set goals, develop better ways to work as a team, and problem-solve; (3) 8 in-home visits in which personal transition trainer/life skills coach provides training, compensatory strategies, and social/technological supports on self-selected activities. The ten visits last 90-120 minutes and ideally take place over a three month period.
  Interventions: Behavioral: Safe@Home Intervention Group
- Usual Care Group (Active Comparator): Participants receive the computer-generated, personalized assessment of abilities, risk, and recommended next steps. Participants may seek services as usual over the 3-month period.
  Interventions: Other: Usual Care Group

INTERVENTIONS:
Behavioral: Safe@Home Intervention Group — For the 8 training visits, participants may select to work on skills in 2 of 5 activity modules: Improving mobility, balance and strength; Managing health and wellness; Staying On Your Own at Home; Maintaining the home; Getting out in the community. Participants may seek single service rehabilitation, medical, and psychological care as usual.
  Arms: Safe@Home Intervention Group
Other: Usual Care Group — Persons can set goals and work on activities with or without a family member as they so choose. Participants may seek single service rehabilitation, medical, and psychological care as usual.
  Arms: Usual Care Group

SUMMARY:
People who sustain moderate to severe traumatic brain injury (TBI) have an increased risk for unintentional injury and harm when resuming day to day activities in the home and community. People who sustain brain injuries primarily want to independently do the activities they enjoy while families primarily focus on avoiding injury or other harm events. Safe@Home is an injury prevention education and activity training program. Participants who have sustained a moderate or severe TBI receive a personalized strengths and safety risk assessment, tailored injury prevention education, and in-home training with a transition coach on self-selected activities. This study will evaluate whether the Safe@Home program reduces injuries and harm and increases clients' independence in their everyday activities in the home and community compared to a usual care control group.

DETAILED DESCRIPTION:
Many persons who have sustained moderate to severe TBI and receive medical rehabilitation transition to their home and community settings with impaired cognition, perceptual motor skills, awareness of disability, self-regulation, and judgment that place them at risk for subsequent unintentional injury or harm. Unintentional injuries often result from falls; motor vehicle or pedestrian events; improper use of electrical equipment, fire, or sharp objects; poisonings; and firearm-related incidents. Risk for harm to self or others also results from victimization, loss of money or valuables, property damage, medication errors, inappropriate responses to emergency or medical situations, and self-regulation problems. Four TBI registry studies have shown that unintentional injury is a leading cause of death (18%-20%) in the year following discharge. In one study, 32% of TBI participants (n=504) had 228 ER visits/hospitalizations from 3-months to several years following discharge due to unintentional injuries.

In order to facilitate independent living and address the safety concerns for persons with TBI in the home and community, a targeted, self-management approach that includes injury prevention education and compensatory strategy training for instrumental activities of daily living (IADLs) is recommended. Institute of Medicine (IOM) and Agency for Healthcare Research and Quality (AHRQ) systematic reviews have recommended the need for TBI post-acute rehabilitation research to find efficient and effective independent living treatments for people with TBI. Rehabilitation investigators recommend evidence-based education that includes integrated, consensus-based, prevention strategies from multidisciplinary rehabilitation professionals to reduce unintentional injury and harm following TBI. Interventions should set goals important to the person with TBI, help the person and family to define roles/responsibilities and work as a team, and develop problem-solving skills and strategies.

The Safe@Home self-management intervention program builds upon our previous research on safety assessment and causes of unsafe events. This clinical trial will evaluate the effectiveness of a person and family-centered intervention to reduce unsafe events and increase self-managed activities and participation. The Safe@Home program is comprised of a personalized assessment report, prevention education and goal-setting, and in-home activity training with a life skills coach. The primary outcomes targeted for this intervention are to: 1) decrease unintentional injury and harm, i.e., unsafe events, and 2) increase independence in daily activities.

Participants will be assigned either to a usual care control group or the Safe@Home program group. Family members of both groups will be asked to complete assessments and both groups of participants and clients and family members will receive a personalized report on their strengths and risks, and suggested strategies to improve independence and reduce risk. The group receiving the Safe@Home Program will also receive in-home education on injury prevention and training on self-selected activities of interest.

Persons with TBI in the Safe@Home program will also be asked to:

* Participate in 2 education sessions to understand their strengths and risks, set goals, work as a team, reduce risks in their home, and problem-solve among themselves, their family member, and personal transition coach
* Participate in 8 in-home visits in which training and supports are provided to help with learning activity skills and compensatory strategies.
* Receive mobile phone and internet reminders to help work on goals and remember strategies.
* Complete a brief questionnaire that should take no longer than 15 minutes before the program, at the end of the program, and 3-months after the program ends.

The questionnaire will ask about:

* their current abilities
* their confidence in their ability to reach goals
* working with their family member on their activity goals and tasks

Family members play an important role in the transition from the hospital to home and have firsthand knowledge of the safety issues that each person with TBI faces.

Family members will be asked to:

* Participate in 2 education sessions to understand the person who had a brain injury strengths and risks, set goals, work as a team, reduce risks in the home, and problem-solve among themselves, their family member who had a brain injury, and personal transition coach
* Complete a questionnaire that should take no longer than 45 minutes to complete before the program, at the end of the program, and 3-months after the program ends.
* Complete a very brief report about unsafe events that should take no longer than 1-2 minutes to complete every 2 weeks.

This questionnaire will ask:

* general background and health information about the family member and the person with TBI
* the likelihood of certain unsafe situations occurring
* the supervision the person with TBI receives
* Mayo-Portland Participation subscale

ELIGIBILITY:
Inclusion Criteria:

Persons with TBI and family members will be eligible if they meet all of the following criteria:

1. Person with TBI aged 18 or older who sustained moderate to severe TBI defined as externally caused damage to brain tissue as evidenced by one of the following (TBI Model Systems Criteria):

   * Post-traumatic Amnesia (PTA) > 24 hours
   * Trauma related intracranial neuroimaging abnormalities
   * Loss of consciousness exceeding 30 minutes (and not due to sedation or intoxication)
   * Glasgow Coma Scale (GCS) score in the emergency department of less than 13 (and not due to intubation, sedation, or intoxication)
2. All participants must be capable of providing informed consent for research participation.
3. Person with TBI has capacity to manage self-care as defined by a rehabilitation specialist rating the patient on the Mayo-Portland Self-Care item ≤ 2, i.e., requires a little assistance or supervision from others, ≤24% of the time.
4. An adult family member, e.g., parent, spouse, adult child, or committed, domestic partner, aged 18 or older, living in the home environment is willing to participate.
5. Person-family resides within 75 miles of the enrollment site and willing to allow a personal transition coach into the home.
6. Person-family willing to use the internet or a mobile phone as part of the intervention.
7. Person-family are English speaking, either native or English as a second language.

Exclusion Criteria:

1. Person with brain injury primary diagnosis is hypoxic or hypoxic-ischemic (i.e., anoxic) brain injury; cerebral infarction (ischemic stroke) or cerebral hemorrhage (i.e., hemorrhagic stroke); intracranial hemorrhage (i.e., aneurismal rupture, subdural or epidural hematoma without TBI); inflammatory, toxic, or metabolic encephalopathies which are not complications of head trauma; seizure disorders (primary generalized epilepsy, partial epilepsies, status epilepticus, etc.); cerebral neoplasm; intracranial surgery; or condition other than moderate or severe TBI as defined above.
2. Person with TBI could not self-manage activities prior to their injury due to severe, uncontrolled psychopathology (e.g., schizophrenia, bipolar disorder) or developmental disability.
3. Person or family has current, severe, untreated/uncontrolled psychopathology (e.g., physically abusive, violent or sexual behavior) that places the personal transition coach treating in the home at physical risk.
4. Person with TBI has severe, current physical or sensory impairment (e.g., tetraplegia, legally blind) that prohibits participation in all activity modules and reflects membership in a different population.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of Unsafe Events for Each Participant | From study start to intervention conclusion (~3-months)
  Actual and near miss unsafe events including injury to self or others, and property damage or loss using a standardized survey
Change in Mayo-Portland Participation Scale Score | Baseline measure and post-intervention measure (~3-months post-baseline)
  Eight items in which amount and level of independence in activities is rated on a 5-point scale

SECONDARY OUTCOMES:
Change in Supervision Rating Scale Score | Baseline, post-intervention (3-months post-baseline), and 3-months post-intervention (6-months post-baseline)
  Amount of supervision provided by a family member on a 13 point scale
Change in Carrying Out Activities Scale Score | Baseline, post-intervention (3-months post-baseline), and 3-months post-intervention (6-months post-baseline)
  Measures level of safety risk associated with cognitive impairment using 17 items rated on a 4-point scale
Number of Unsafe Events for Each Participant | From intervention conclusion to 3-months post-intervention
  Actual and near miss unsafe events including injury to self or others, and property damage or loss using a standardized survey
Change in Mayo-Portland Participation Scale Score | Baseline measure and 3-month post-intervention measure (6-months post-baseline)
  Eight items in which amount and level of independence in activities is rated on a 5-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T. Seel, PhD, Principal Investigator — Shepherd Center, Atlanta GA
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The principal investigator will ensure that all data sharing requirements of the funding agency are met. There is not a formal plan for sharing data at this time.